CLINICAL TRIAL: NCT04548999
Title: A Phase IIIB Multicenter, Randomized, Double-blind, Controlled Study to Evaluate the Efficacy, Safety and Pharmacokinetics of a Higher Dose of Ocrelizumab in Adults With Primary Progressive Multiple Sclerosis
Brief Title: A Study to Evaluate the Efficacy, Safety and Pharmacokinetics (PK) of a Higher Dose of Ocrelizumab in Adults With Primary Progressive Multiple Sclerosis (PPMS)
Acronym: GAVOTTE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN42083; 2020-000894-26 (EudraCT Number); 2023-506515-18-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Primary Progressive Multiple Sclerosis; Higher Dose of CD20 Antibody Ocrelizumab; Efficacy, Safety and Pharmacokinetics
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — ocrelizumab; Histamine Antagonists; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab Higher Dose (Experimental): Participants will be randomized to receive a minimum of 5 higher treatment doses based on their body weight at baseline: 1200 mg (participant's body weight <75 kilograms [kg]) or 1800 mg (participant's body weight ≥ 75 kg) of ocrelizumab administered by IV infusion Q24W in the DBT phase. During the optional OLE phase, participants will continue with their assigned dose of ocrelizumab (either 1200 or 1800 mg) for approximately 96 weeks (4 doses in total). Mandatory methylprednisolone (or equivalent) and antihistaminic drug (e.g., diphenhydramine or equivalent) will be administered approximately 30-60 minutes prior to the start of each ocrelizumab infusion.
  Interventions: Drug: Ocrelizumab; Drug: Antihistamine; Drug: Methylprednisolone
- Ocrelizumab Approved Dose (Active Comparator): Participants will be randomized to receive a minimum of 5 treatment doses of 600 mg ocrelizumab administered by IV infusion Q24W in the DBT phase. During the optional OLE phase, participants will be offered a higher dose of ocrelizumab (either 1200 or 1800 mg), based on their body weight at OLE baseline, for approximately 96 weeks (4 doses in total). Mandatory methylprednisolone (or equivalent) and antihistaminic drug (e.g., diphenhydramine or equivalent) will be administered approximately 30-60 minutes prior to the start of each ocrelizumab infusion.
  Interventions: Drug: Ocrelizumab; Drug: Antihistamine; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Ocrelizumab — The actual higher dose of ocrelizumab will be assigned to participants based on their body weight at baseline: 1200 mg (body weight <75 kg) or 1800 mg (body weight ≥ 75 kg). The first dose of ocrelizumab will be administered as two 600 mg or 900 mg IV infusions given 14 days apart. For the subsequent doses, ocrelizumab will be administered as a single 1200 mg or 1800 mg IV infusion Q24W.
  During the optional OLE phase, participants will continue with their assigned dose of ocrelizumab (either 1200 or 1800 mg) for approximately 96 weeks (4 doses in total)
  Other Names: Ocrevus
  Arms: Ocrelizumab Higher Dose
Drug: Ocrelizumab — Ocrelizumab will be administered at a dose of 600 mg Q24W. The first dose of ocrelizumab will be administered as two 300 mg, IV infusions given 14 days apart. For the subsequent doses, ocrelizumab will be administered as a single 600 mg IV infusion Q24W.
  Other Names: Ocrevus
  Arms: Ocrelizumab Approved Dose
Drug: Antihistamine — Premedication with oral or IV antihistaminic drug (i.e., diphenhydramine 50 mg or an equivalent dose of an alternative) will be administered prior to each ocrelizumab infusion.
  Other Names: Non-Investigational Medicinal Product
Drug: Methylprednisolone — Premedication with 100 mg of methylprednisolone (or equivalent) will be administered by IV infusion prior to each ocrelizumab infusion.
  Other Names: Non-Investigational Medicinal Product

SUMMARY:
This is a randomized, double blind, controlled, parallel group, multicenter study to evaluate efficacy, safety and PK of a higher dose of ocrelizumab per intravenous (IV) infusion every 24 weeks (Q24W) in participants with PPMS, in comparison to the approved 600 milligrams (mg) dose of ocrelizumab.

DETAILED DESCRIPTION:
Participants will be treated for a minimum of 120 weeks in the double-blind treatment (DBT) phase. Upon positive primary results after the DBT phase, an optional higher dose extension treatment, open-label extension (OLE) phase is planned for eligible participants. The OLE will be carried out for approximately 96 weeks. Participants will be followed for safety for 48 weeks thereafter. Participants whose B-cell levels still did not replete to their baseline level or the lower limit of normal (LLN), whichever is lower, will move into the B-cell monitoring (BCM) phase following the safety follow-up phase. The study will end when all participants who were not treated with an alternative B-cell depleting therapy have repleted their B-cells to the baseline value or the LLN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPMS
* EDSS score at screening and baseline, from 3 to 6.5 inclusive
* Average T25FWT score over two trials at screening and over two trials at baseline respectively, up to 150 (inclusive) seconds
* Average 9HPT score over four trials (two trials with each hand) at screening and over four trials (two trials with each hand) at baseline respectively, up to 250 (inclusive) seconds
* Score of ≥ to 2.0 on the Functional Systems (FS) scale for the pyramidal system that was due to lower extremity findings at screening and baseline
* Documented magnetic resonance imaging (MRI) of brain with abnormalities consistent with MS
* Participants requiring symptomatic treatment for MS and/or physiotherapy must be treated at a stable dose. No initiation of symptomatic treatment for MS or physiotherapy within 4 weeks of randomization
* Participants must be neurologically stable for at least 30 days prior to randomization and baseline
* Disease duration from the onset of MS symptoms; if EDSS score at screening is ≤ 5, disease duration must be less than 10 years; If EDSS score at screening is > 5, disease duration must be less than 15 years
* Documented evidence of the presence of at least one cerebrospinal fluid-specific oligoclonal bands
* Females of childbearing potential: agreement to remain abstinent or use adequate contraceptive methods
* Female participants, without reproductive potential may be enrolled e.g. if post-menopausal or if surgically sterile

Exclusion Criteria:

* History of relapsing remitting or secondary progressive MS at screening
* Any known or suspected active infection at screening or baseline (except nailbed infections), or any major episode of infection requiring hospitalization or treatment with IV antimicrobials within 8 weeks or treatment with oral antimicrobials within 2 weeks, prior to and during screening
* History of confirmed or suspected progressive multifocal leukoencephalopathy
* History of cancer, including hematologic malignancy and solid tumors, within 10 years of screening
* Immunocompromised state
* Receipt of a live or live-attenuated vaccine within 6 weeks prior to randomization
* Inability to complete an MRI or contraindication to gadolinium administration
* Contraindications to mandatory pre-medications for infusion-related reaction (IRRs)
* Known presence of other neurologic disorders that could interfere with the diagnosis of MS or assessments of efficacy and/or safety during the study
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* Significant, uncontrolled disease that may preclude participant from participating in the study
* History of or currently active primary or secondary, non-drug-related, immunodeficiency
* Pregnant or breastfeeding or intending to become pregnant
* Lack of peripheral venous access
* History of alcohol or other drug abuse within 12 months prior to screening
* Treatment with any investigational agent or treatment with any experimental procedure for MS
* Previous use of anti-cluster of differentiation 20 (CD20s) (including ocrelizumab), unless the last infusion was more than 2 years before screening, B-cell count is normal, and the stop of the treatment was not motivated by safety reasons or lack of efficacy
* Any previous treatment with mitoxantrone, cladribine, atacicept, alemtuzumab, and daclizumab
* Previous treatment with fingolimod, siponimod, or ozanimod within 6 weeks of baseline
* Previous treatment with natalizumab within 4.5 months of baseline
* Previous treatment with interferons beta (1a or 1b), or glatiramer acetate within 2 weeks of baseline
* Previous treatment with any other immunomodulatory or immunosuppressive medication not already listed above without appropriate washout as described in the applicable local label. If the washout requirements are not described in the applicable local label, then the wash out period must be five times the half-life of the medication
* Any previous treatment with bone marrow transplantation and hematopoietic stem cell transplantation
* Any previous history of transplantation or anti-rejection therapy
* Treatment with IV immunoglobulin (Ig) or plasmapheresis within 12 weeks prior to randomization
* Systemic corticosteroid therapy within 4 weeks prior to screening
* Positive screening tests for active, latent, or inadequately treated hepatitis B
* Sensitivity or intolerance to any ingredient (including excipients) of ocrelizumab
* Any additional exclusionary criterion as per ocrelizumab local label, if more stringent than the above

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 769 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2027-09-08 (Estimated)

PRIMARY OUTCOMES:
Time to Onset of Composite Confirmed Disability Progression (cCDP) Sustained for at least 12 Weeks | Baseline up to approximately 4.3 years
  Time to onset of cCDP is defined as the first occurrence of a predefined confirmed progression event measured by Expanded Disability Status Scale (EDSS), Timed 25-foot Walk Test (T25FWT) or 9-hole Peg Test (9-HPT)

SECONDARY OUTCOMES:
Time to Onset of 12-week Composite Confirmed Disability Progression (cCDP12) Independent of Protocol-defined Relapses (PDR) | Baseline up to approximately 4.3 years
  Time to onset of cCDP is defined as the first occurrence of a predefined confirmed progression event measured by EDSS, T25FWT or 9-HPT independent of PDR
Time to Onset of 12-week Confirmed Disability Progression (CDP12) | Baseline up to approximately 4.3 years
  CDP, defined as a sustained increase from baseline in EDSS score of ≥1.0 point in participants with a baseline EDSS score of ≤5.5 or a sustained increase of ≥0.5 points in participants with a baseline EDSS score of >5.5
Time to ≥ 20% Increase in 12-week Confirmed by T25FWT | Baseline up to approximately 4.3 years
  The T25FWT is a performance measure used to assess walking speed based on a timed 25-foot walk. The participant is directed to start at one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly and safely as possible.
Change in Neurofilament Light (NfL) at Week 96 | Baseline up to Week 96
  Biomarker for neurodegeneration NfL
Time to 12-week Confirmed 8-point Increase in 12-item Multiple Sclerosis Walking Scale (MSWS12) | Baseline up to approximately 4.3 years
  Self-reported measure of the impact of multiple sclerosis (MS) on the individual's ability to walk
Annual Rate of Percent Change From Baseline in Total Brain Volume | Baseline up to approximately 4.3 years
Annual Rate of Percent Change From Baseline in Thalamic Volume | Baseline up to approximately 4.3 years
Time to 12-week Confirmed 4-point Worsening in Symbol Digit Modality Test (SDMT) | Baseline up to approximately 4.3 years
  The SDMT is a performance measure that has demonstrated sensitivity in detecting not only the presence of cognitive impairment but also changes in cognitive functioning over time and in response to treatment. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Responses will be collected orally. A four-point change from baseline is typically considered clinically meaningful.
Change in NfL (i.e. Ratio to Baseline) at Week 96 for Participants in the Approved Dose Ocrelizumab Group | Baseline up to Week 96
  Biomarker for neurodegeneration NfL
Change in NfL (i.e. Ratio to Baseline) at Week 96 for Participants in the Higher Dose Ocrelizumab Group | Baseline up to Week 96
  Biomarker for neurodegeneration NfL
Time to Onset of 24-week Composite Confirmed Disability Progression (cCDP24) Independent of PDR | Baseline up to approximately 4.3 years
  Time to onset of cCDP is defined as the first occurrence of a predefined confirmed progression event measured by EDSS, T25FWT or 9-HPT independent of PDR
Percentage of Participants With Adverse Events (AEs) | Baseline up to approximately 8 years
Serum Concentrations of Ocrelizumab at Specified Timepoints | Weeks 0, 2, 12, 24, 36, 48, 60, 72, 84, 96, 120
Change in B-cell Levels in Blood | Baseline up to approximately 4.3 years
Percentage of Participants Achieving 5 or Less B-cells per Microliter of Blood | Baseline up to approximately 4.3 years
Change From Baseline in the Anti-drug Antibody (ADA) Levels | Week 0, 24, 48, 72, 96, 120

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (149):
- United States (24):
  - Alabama Neurology Associates, Homewood, Alabama
  - 21st Century Neurology, Phoenix, Arizona
  - University of California Irvine, Irvine, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Advanced Neurosciences Research LLC, Fort Collins, Colorado
  - MS and Neuromuscular Center of Excellence, Clearwater, Florida
  - University of South Florida, Tampa, Florida
  - Baptist Health Lexington, Nicholasville, Kentucky
  - International Neurorehabilitation Institute, Lutherville, Maryland
  - Massachusetts General Hospital., Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Jersey Shore University Medical Centre, Neptune City, New Jersey
  - Northwell Health, Great Neck, New York
  - Lenox Hill Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Neurology Clinic PC, Cordova, Tennessee
  - Advanced Neurosciences Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Lone Star Neurology of San Antonio, San Antonio, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - Wheaton Franciscan Healthcare - St. Francis Outpatient Center, Milwaukee, Wisconsin
- Argentina (3):
  - CEMIC Saavedra, Buenos Aires
  - Centro de Especialidades Neurológicas y Rehabilitación - CENyR, Buenos Aires
  - INECO, Rosario
- Revalidatie en MS Centrum, Overpelt, Belgium
- Brazil (11):
  - L2 Ip Instituto de Pesquisas Clinicas Ltda ME, Brasília, Federal District
  - Hospital das Clinicas - UFG, Goiânia, Goiás
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - IMV Pesquisa Neurológica, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Clinica Neurologica, Joinville, Santa Catarina
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Praxis Pesquisa Médica, Santo André, São Paulo
  - CPQuali Pesquisa Clinica Ltda, São Paulo, São Paulo
- Bulgaria (2):
  - UMHAT Dr. Georgi Stranski, Pleven
  - MHATNP Sveti Naum EAD, Sofia
- Canada (3):
  - Centre de Recherche Saint-Louis, Lévis, Quebec
  - Chum Campus Notre Dame, Montreal, Quebec
  - MUCH - Montreal Neurological Institute & Hospital, Montreal, Quebec
- Denmark (2):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet Glostrup, Glostrup Municipality
- France (7):
  - CHU de Besancon Hopital Jean Minjoz, Besançon
  - CHU Brest Hopital La Cavale Blanche, Brest
  - Hopital Cote De Nacre, Caen
  - CHU Hopital Gabriel Montpied, Clermont-Ferrand
  - CH St Vincent de Paul, Lille
  - Hopital Central - CHU de Nancy, Nancy
  - Hopital Hautepierre - CHU Strasbourg, Strasbourg
- Germany (8):
  - Universitätsklinikum "Carl Gustav Carus", Zentrum für Klinische Neurowissenschaften, Dresden
  - Universitätsmedizin Greifswald, Greifswald
  - Medizinische Hochschule Hannover, Klinik für Neurologie, Hanover
  - Universität Leipzig, Leipzig
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Deutsche Klinik für Diagnostik, Wiesbaden
- Greece (2):
  - Hospital Eginition, Athens
  - 401 Military Hospital of Athens, Athens
- Hungary (5):
  - Semmelweis Egyetem Idegsebeszeti és Neurointervencios Klinika, Budapest
  - UNO Medical Trials Kft., Budapest
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
- Italy (7):
  - A. O. U. Federico II, Napoli, Campania
  - AOU Seconda Università degli Studi, Napoli, Campania
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Ospedale S.Antonio Abate, Gallarate, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - IRCCS Istituto Neurologico C. Mondino?Dip. Neurologia Neuroriabilitazione S.S. Sclerosi Multipla, Pavia, Lombardy
  - AOU Città della Salute e della Scienza, Turin, Piedmont
- Mexico (4):
  - Centro de Investigacion Medico Biologico y Terapia Avanzada, S.C., Guadalajara, Jalisco
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - Neurociencias Prisma, A.C, San Luis Potosí City, San Luis Potosí
  - Grupo Médico Camino S.C., México
- Peru (3):
  - Hospital Nacional Guillermo Almenara Irigoyen, La Victoria, Lima
  - Instituto Nacional de Ciencias Neurológicas - Hospital Mogrovejo, Lima
  - Hospital Nacional Dos de Mayo, Lima
- Poland (14):
  - Neurocentrum Bydgoszcz sp. z o.o, Bydgoszcz
  - COPERNICUS Podmiot Leczniczy Sp. z o. o. Szpital im. M. Kopernika, Gdansk
  - MA-LEK Clinical Sp. Z o.o., Katowice
  - Szpital Specjalistyczny im. Rydygiera w Krakowie, Krakow
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Indywidualna Praktyka Lekarska Prof. Dr Hab. N. Med. Konrad Rejdak., Lublin
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. z o.o. Sp. k., Oświęcim
  - Neurologiczny Niepubliczny ZOZ Centrum Leczenia SM Osrodek Bada? Klinicznych, Plewiska
  - EMC Instytut Medyczny SA, Późna
  - Wojewódzki Szpital Specjalistyczny Nr 3, Rybnik
  - Nmedis sp. z o.o., Rzeszów
  - Osrodek Badan Klinicznych Euromedis, Szczecin
  - Centrum Medyczne NeuroProtect, Warsaw
  - Instytut Psychiatrii i Neurologii II Klinika Neurologiczna, Warsaw
- Portugal (4):
  - Hospital de Braga, Braga
  - Hospital Santo Antonio dos Capuchos, Lisbon
  - Centro Hospitalar de Lisboa Ocidental - Hospital Egas Moniz, Lisbon
  - Hospital Geral de Santo Antonio, Porto
- Russia (16):
  - Krasnoyarsk State Medical Academy, Krasnoyarsk, Krasnoyarsk Krai
  - FSBHI Siberian Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk, Krasnoyarsk Krai
  - Research Center of Neurology of RAMS, Moscow, Moscow Oblast
  - Federal center of brain research and neurotechnologies, Moskva, Moscow Oblast
  - City Clinical Hospital #24, Moskva, Moscow Oblast
  - Leningrad Regional Clinical Hospital, Saint Petersburg, Sankt-Peterburg
  - National Center of Social Significant Disease, Saint Petersburg, Sankt-Peterburg
  - N.P. Bechtereva Institute of the Human Brain, Saint Petersburg, Sankt-Peterburg
  - City Hospital #40 of Kurortniy Administrative District, Saint Petersburg, Sankt-Peterburg
  - SHI Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg, Sverdlovsk Oblast
  - Vertebronevrologiya LLC, Kazan', Tatarstan Republic
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk, Ulyanovsk Oblast
  - Center of Cardiology and Neurology, Kirov
  - Regional clinical hospital named after prof. S.V. Ochapovsky, Krasnodar
  - FSBIH Siberian Regional Medical Centre of FMBA of Russia, Novosibirsk
  - Perm SMA n.a. academ. E.A. Vagner, Perm
- Spain (4):
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta De Hierro Majadahonda, Madrid
  - Hospital Universitario Virgen de Arrixaca, Murcia
- Inselspital Bern Medizin Neurologie, Bern, Switzerland
- Turkey (Türkiye) (12):
  - Gazi University Medical Faculty, Ankara
  - Baskent Universitesi Ankara Hastanesi, Çankaya
  - Haseki Training and Research Hospital, Istanbul
  - Istanbul Universitesi - Cerrahpasa Cerrahpasa Tip Fakultesi, Istanbul
  - Sancaktepe Training and Research Hospital, Istanbul
  - Selcuk University Medical Faculty, Istanbul
  - Erciyes Universitesi, Kayseri
  - Kocaeli University Hospital, Kocaeli
  - Ege Üniversitesi Tip Fakültesi, Lzmir
  - Cumhuriyet Universitesi Tip Fakultesi, Merkez
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis University School of Medicine, Samsun
- Ukraine (12):
  - 5th Cherkasy City Center of Primary Health Care, Cherkasy
  - SI USSRI of Medical and Social Problems of Disabilities of MOHU, Dnipro
  - Regional Clinical Hospital, Ivano-Frankivsk
  - St.In.Inst. of Neurol.Psych.and Narcol.of the AMSU, Kharkiv
  - State Institution Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine, Kharkiv
  - Medical Center Dopomoga Plus, Kyiv
  - Medical Center of Private Execution First Private Clinic, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Lvivska oblasna tsentralna likarnia, Lviv
  - Sumy Regional Clinical Hospital, Sumy
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsi
  - Municipal Non-profit Enterprise Zaporizhzhya Regional Hospital Zaporizhzhya Regional Council, Zaporizhzhia
- United Kingdom (4):
  - Charing Cross Hospital, London
  - National Hospital for Neurology and Neurosurgery,, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing